CLINICAL TRIAL: NCT05648409
Title: Comparison of the Body Mass Index, Visceral Adiposity Index, the Body Shape Index, and the Body Roundness Index With the Metabolic Score for Visceral Adiposity in the Assessment of Visceral Adiposity
Brief Title: Comparison of Body Mass Index and Metabolic Score for Visceral Adiposity in Evaluation of Visceral Adiposity
Status: Completed | Type: Observational
Sponsor: Goztepe Prof Dr Suleyman Yalcın City Hospital (Other)
Responsible Party: Principal Investigator, Cundullah Torun, Principal Investigator, Goztepe Prof Dr Suleyman Yalcın City Hospital
Other Study IDs: METSVF-adiposity
Record Dates: First submitted 2022-11-15; First posted 2022-12-13 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Visceral Obesity
Keywords: visceral adiposity; metabolic score for visceral fat (METS-VF); body mass index
MeSH Terms: conditions — Obesity, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Visceral obesity is a major risk factor for cardiometabolic diseases such as type 2 diabetes, hypertension, and coronary artery disease. In clinical settings and during research, "body mass index (BMI)" is usually used for assessing obesity, and when it is above 30 kg/m2, it is defined as obesity. However, the risk posed by obesity is more related to body fat distribution than total body fat, and BMI only reflects the second. Individuals with a BMI below 30, even 25, may still have visceral adiposity detectable via an abdominal computerized tomography ( CT) or magnetic resonance imaging (MRI). Therefore new, practical, inexpensive parameters are needed to evaluate visceral adiposity. "Metabolic Score for Visceral Adiposity (METS-VF)", "Body Shape Index (BSI)", "Conicity Index (CI)" and "Body Roundness Index (BRI)" are a few recent indexes developed trying to fulfill these needs. The aim is to investigate the effectivity of METS-VF in comparison with BMI, BSI, CI, and BRI in reflecting visceral adiposity assessed with CT.

DETAILED DESCRIPTION:
This study is a single-center, observational and prospective study. Patients who underwent abdominal computed tomography (CT) covering the L3-L4 level in the last month for any reason and who did not have any of the following situations in the participants' CT reports: malignancy, pancreatitis, diseases requiring further investigation, chronic inflammatory diseases, and a pathology requiring hospitalization for more than 24 hours, will be invited to the study. Of the patients who consent to the study, gender, age, education level, current diseases, medications, and smoking status are questioned. Anthropometric measurements, especially waist, height, and weight are taken. Patients' biochemical parameters such as lipid profiles (LDL-cholesterol, HDL-cholesterol, Triglyceride), urea, creatinine, uric acid, fasting blood glucose, and C-peptide levels (after 8-12 hours of fasting), and thyroid hormones were measured in the last three months are recorded from the participants' files. The body mass index (BMI) of the patients will be calculated with the formula weight (kg) / height (m)2. Patients will be in 5 groups with BMI <25 kg/m2, 25-29.9 kg/m2, 30-34.9 kg/m2, 35-39.9 kg/m2, and >40 kg/m2, with 40 patients in each group. Visceral adipose tissue will be calculated by the radiologist by measuring with the "slicer" method at the level of L3-4 on abdominal CT. For "Metabolic Score for Visceral Fat (METS-VF)", the formula 4.466 + 0.011*(Ln(METS-IR))3 + 3.239*(Ln(Waist/height ratio))3 + 0.319*(Gender) + 0.594*(Ln(Age)) and for "Body Waist Circumference" the formula (BMI2/3 * height1/2) are used. Based on the visceral adipose tissue measured by CT, firstly, BMI and METS-VF will be compared, and then the other mentioned anthropometric index values will be compared statistically. The assumption is that the METS-VF index is superior to the other indexes, including the BMI. Also, as a second endpoint, it is aimed to find a cut-off value for METS-VF in Turkish individuals to reflect the increased visceral adiposity assessed with CT.

ELIGIBILITY:
Inclusion Criteria:

* Having consented to the work
* Having a computed tomography of the abdomen taken within the last month
* Having a biochemistry analysis including lipid levels in the last three months
* No weight loss in the last 3 months

Exclusion Criteria:

* Antihyperlipidemic medication usage
* Presence of active malignancy
* Having an anatomical structure that is not suitable for taking anthropometric measurements
* The use medications that might affect metabolic values such as steroids
* Chronic inflammatory diseases, acute infection and other lipodystrophic syndromes (HIV etc.)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients aged between 20 and 50 years old who underwent abdominal computed tomography (CT) imaging, including the L3-L4 level for any reason in the last month, with no detectable malignancy, pancreatitis, diseases requiring further investigation, chronic inflammatory diseases, and a pathology necessitating hospitalization for more than 24 hours in the CT evaluation, we're invited to the study.
Sampling Method: Non-Probability Sample
Enrollment: 194 (Actual)
Dates: Start 2022-01-10 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
The Superiority of the Metabolic Score for Visceral Fat (METS-VF) on the Body Mass Index (BMI) for visceral adiposity | through study completion, an average of 1 year
  The study aims to evaluate the effectiveness of the Metabolic Score for Visceral Fat (METS-VF) on the evaluation of visceral adiposity compared with the Body Mass Index (BMI). For METS-VF, a cut-off value will be determined. For BMI values 20-24.9 are accepted as normal, 25-29.9 as overweight and above 30 as obese (with different categories), whereas below 20 as underweight.
The Superiority of the Metabolic Score for Visceral Fat (METS-VF) on the Visceral Adiposity Index (VAI) for visceral adiposity | through study completion, an average of 1 year
  The number of participants whose visceral adiposity, which was evaluated by abdominal computerized tomography, was correctly assessed by using the Metabolic Score for Visceral Fat (METS-VF) and Visceral Adiposity Index (VAI) for which higher values are predicted to reflect higher adiposity.
The Superiority of the Metabolic Score for Visceral Fat (METS-VF) on the Body Shape Index (ABSI) for visceral adiposity | through study completion, an average of 1 year
  The number of participants whose visceral adiposity, which was evaluated by abdominal computerized tomography, was correctly assessed by using the Metabolic Score for Visceral Fat (METS-VF) and the Body Shape Index (ABSI) for which higher values are predicted to reflect higher adiposity.
The Superiority of the Metabolic Score for Visceral Fat (METS-VF) on the Body Roundness Index (BRI) for visceral adiposity | through study completion, an average of 1 year
  The number of participants whose visceral adiposity, which was evaluated by abdominal computerized tomography, was correctly assessed by using the Metabolic Score for Visceral Fat (METS-VF) and the Body Roundness Index (BRI) for which higher values are predicted to reflect higher adiposity.
The Superiority of the Metabolic Score for Visceral Fat (METS-VF) on the evaluation of visceral adiposity | through study completion, an average of 1 year
  The number of participants whose visceral adiposity, which was evaluated by abdominal computerized tomography, was correctly assessed by using the Metabolic Score for Visceral Fat (METS-VF) and the other defined indexes, the Body Mass Index (BMI), Visceral Adiposity Index (VAI), the Body Shape Index (ABSI), and the Body Roundness Index (BRI) with the purpose of finding the best discriminator for visceral adiposity.

SECONDARY OUTCOMES:
Determination of a cut-off point for METS-VF score associated with increased Visceral Adiposity | through study completion, an average of 1 year
  Using receiver-operating characteristics (ROC) curve analysis with the calculated input from the abdominal computerized tomography and the Metabolic Score for Visceral Fat (METS-VF) index. METS-VF index is a continuous index with no definite cut-off value. For different populations a new cut-off point is calculated, which it is also aimed in this study. The higher the score, the higher is the expected visceral adiposity.

CONTACTS AND LOCATIONS:
Overall Officials: Cundullah Torun, MD, Principal Investigator — Istanbul Goztepe Prof Dr Suleyman Yalcin City Hospital, Egitim mah. Kadıköy/ İstanbul, TURKEY
Locations (1):
- Istanbul Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Torun C, Ankarali H, Castur L, Uzunlulu M, Erbakan AN, Akbas MM, Gunduz N, Dogan MB, Oguz A. Is Metabolic Score for Visceral Fat (METS-VF) a Better Index Than Other Adiposity Indices for the Prediction of Visceral Adiposity. Diabetes Metab Syndr Obes. 2023 Aug 29;16:2605-2615. doi: 10.2147/DMSO.S421623. eCollection 2023. PMID 37663201